CLINICAL TRIAL: NCT05921357
Title: Evaluation of Fermented Foods and Probiotic Consumption Frequency in Peri-implant Disease and Health
Brief Title: Effect of Fermented Products and Probiotics on the Condition of the Implant
Acronym: EFFPCFPDH
Status: Completed | Type: Observational
Sponsor: Tuğba ŞAHİN (Other)
Responsible Party: Sponsor-Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Organization: Abant Izzet Baysal University (Other)
Other Study IDs: 2022/196
Record Dates: First submitted 2023-06-18; First posted 2023-06-27 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Implant
Keywords: Fermented foods; probiotics; peri-implant health; peri-implant mucositis; peri-implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Peri-implantitis: Implants with a pocket depth of more than 5 mm and bleeding on probing
  Interventions: Other: Questionnaire
- Peri-implant mucositis: Implants with no bone loss but bleeding on probing
  Interventions: Other: Questionnaire
- Peri-implant health: Implants with no bone loss but no bleeding on probing
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire and examine

SUMMARY:
126 individuals with peri-implant disease and health, aged between 18-70 years, who applied to Bolu University Faculty of Dentistry Periodontology Clinic, participated in the study.The inclusion criteria for patient participation in the study were: age of patients between 18 and 70 years; the presence of at least 20 natural teeth in the oral cavity; systemic health. Peri-implant status was determined by the clinician (T.Ş.) by evaluating dental implants' plaque, gingival index, bleeding on probing, pocket depth measurements, and clinical attachment level. In addition, them systemic illness, pregnancy, breastfeeding status, medication, antibiotic use, and whether they smoked were questioned. Systemically unhealthy patients who did not use antibiotics within a month, were breastfeeding or pregnant, had uncontrolled diabetes, rheumatic fever, a history of lung and kidney disorders, and used drugs that could affect periodontal tissues were not included in the study. After examination, the patients were divided into three groups according to their disease: Peri-implantitis (42 patients), peri-implantitis (42 patients), and peri-implant health (42 patients). Demographic characteristics (age, weight, gender, height, education, and employment status) of the participants were collected with a questionnaire. With this survey, fermented foods and probiotic products such as bacon, soy sauce, pickles, sourdough bread, whole grain, rye, wholemeal bread, ayran, kefir, turnip, vinegar (homemade), pomegranate syrup (homemade), probiotic beverage, the frequency and amount of consumption of cheese, dark chocolate, tablets, capsules, chassis, butter and other (Kimchi, sauerkrauth, miso soup, fermented herring, kombucha, etc.) were determined. It was requested to determine the relationship between the health and disease of the implant and the frequency of consumption of fermented and probiotic products and foods in individuals with implants.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals
* Individuals between the ages of 18-70

Exclusion Criteria:

* No use of antibiotics within one month
* Breastfeeding or being pregnant
* Uncontrolled diabetes, rheumatic fever, history of lung and kidney disorders, and drug use that will affect periodontal tissues

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bolu Abant İzzet Baysal University
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Consumption frequency | Baseline
  the number of times a product is consumed in a given time period.
Consumption amount | Baseline
  The average quantity of an item consumed or expended during a given time interval, expressed in quantities by the most appropriate unit of measurement per applicable stated basis.
Daily intake | Baseline
  The amount of a substance that people can consume on a daily basis
Bleeding on probing | Baseline
  Bleeding, leading sign of inflammation inside the connective tissue, is a critical factor for pocket depth measurements, and with other variable factors prevents making reproducible measurements.
Periodontal pocket depth | Baseline
  a pathologically deepened gingival sulcus around a tooth at the gingival margin.

SECONDARY OUTCOMES:
Plaque index | Baseline
  The plaque index assesses the amount of dental plaque visible on the vestibular and lingual surfaces of all teeth
Gingival index | Baseline
  This measurement is based on the presence or absence of bleeding on gentle probing.
Clinical attachment level | Baseline
  CAL is calculated by subtracting the gingival margin level from the probing depth.

CONTACTS AND LOCATIONS:
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided